CLINICAL TRIAL: NCT03004079
Title: Assessment of the Clinical Importance of Insulin Resistance & Steroid-Associated Hyperglycemia in Relapsing Multiple Sclerosis
Brief Title: Clinical Importance of Glucose Regulation in Relapsing MS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Myla Goldman, MD, Associate Professor of the Department of Neurology, University of Virginia
Other Study IDs: 19259
Record Dates: First submitted 2016-11-02; First posted 2016-12-28 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the relationship of blood glucose levels in persons with Multiple Sclerosis (MS) who have experienced a relapse and will be receiving intravenous steroids for the relapse, to their recovery from the relapse.

Steroid exposure commonly leads to elevated serum blood glucose, however, standardized monitoring of blood glucose levels in the outpatient setting is not common. The clinical impact of any associated elevated blood glucose during steroid administration is unknown. We hypothesize that the blood glucose response to steroid treatment is clinically relevant to the MS-relapse recovery.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a neuroinflammatory and degenerative central nervous system disorder. The majority of patients have an early relapsing-remitting course. Standard treatment for an MS-relapse is intravenous methylprednisolone (IVMP), typically 1000 mg daily for 3 days. Despite IVMP treatment, >40% of MS patients experience residual deficits after an MS-relapse. Potential risk factors for poor relapse recovery remain unclear.

Elevated serum blood glucose is a common and well-defined consequence of steroid administration, attributed to steroid-related reductions in insulin sensitivity. Individuals with pre-treatment insulin resistance (e.g. diabetics) will exhibit an amplified hyperglycemic response. Reduced mobility, sedentary lifestyle, and repeated exposure to steroids- all of which are common in MS - are recognized risk factors for insulin resistance. These factors may make MS patients particularly susceptible to steroid-induced hyperglycemia. While, MS patients commonly receive intravenous steroids, the clinical impact of any associated hyperglycemia is unknown.

Study Design and Methods Timeline: Study will require 3 visits over a 6 month period.

Subjects: MS subjects who are experiencing an acute relapse will be recruited for the study. Prior to any study procedures, the PI or research coordinator will obtain full written informed consent.

Baseline Measurements: age, race/ethnicity, sex, weight, height, waist circumference, blood pressure, previous steroid exposure (dates, frequency, steroid type and dose), smoking history, and family history of diabetes. Medication review will include MS disease-modifying therapy, symptomatic medications, and non-MS-related medications. Additional MS-related information will include dates of initial MS-symptom onset, MS diagnosis, and onset of presenting relapse symptoms.

Oral glucose tolerance test (OGTT) & Matsuda Index: Prior to steroid administration, MS subjects will undergo a 2-hour OGTT. OGTT and Matsuda Index will then be repeated at the 3- and 6-month follow-up visits.

Blood studies: HgA1c (hemoglobin A1C), a fasting lipid panel (LDL-C, HDL-C, triglycerides, and total cholesterol), insulin growth factor, vitamin D level, adiponectin level, homocysteine level, and leptin level. All laboratory tests completed at baseline, 3- and 6-month visits.

Surveys: Subjects will complete surveys related to their perceived disability, relapse severity and recovery, and other MS-related symptoms.

Functional testing: EDSS, MS Functional Composite, timed-walk testing, accelerometry, low contrast visual acuity test (LCVA) and the symbol digit modality test (SDMT).

Intravenous steroid treatment: Standardized 1000 mg of intravenous methylprednisolone (IVMP) daily for 3 days (reconstituted in 0.9% sodium chloride). IVMP will be billed to patient insurance as part of routine clinical care.

Blood glucose monitoring: Bayer Contour Next glucometer will be used to measure capillary BG levels 6 times daily (Subjects will be instructed to check their BG starting on the day of screening and to continue BG checks (as above) until their return appointment 5-7 days after steroid treatment completion for a total of 8-10 days. Subjects will be required to avoid snacks between meals for the 3 days of IVMP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Age 18 -59 years (inclusive)
* Ability to walk continuously for 6 minutes (per patient report)
* Clinically Isolated Syndrome (CIS) or Relapsing Remitting MS (RRMS) confirmed diagnosis by McDonald 2010 criteria

  * Current MS relapse with objective findings on exam
  * Relapse symptom onset within 2-weeks of screening
  * Functional System Scores obtainable from a clinic visit within 6 months of the relapse assessment visit
  * EDSS < 6.5 at time of screening visit
  * Inpatient, outpatient, emergency department, or inpatient observation status

Exclusion Criteria:

* Prior steroid exposure within 90 days of enrollment
* HgA1c ≥ 6.5 at baseline screening
* Evidence of concurrent infection
* Known contraindications to IV steroid treatment
* History of diabetes mellitus ( type 1 or 2) or severe hypertension
* Use of any glucose-regulating medications
* Pregnancy or current use of hormone replacement therapy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 18-54 (inclusive) with a diagnosis of clinically isolated syndrome or relapsing remitting multiple sclerosis with an acute attack (relapse).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Relapse Recovery & Hyperglycemia | Recovery from relapse at 6-months
  Determine the relationship between mean postprandial blood glucoses (BG) and relapse recovery (complete vs. incomplete) following a standardized IVMP treatment.
Insulin Resistance & Relapse Severity | At Baseline
  Determine if insulin resistance (IR), measured by the Matsuda Index, is an independent predictor of relapse severity.

CONTACTS AND LOCATIONS:
Overall Officials: Myla Goldman, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nickerson M, Marrie RA. The multiple sclerosis relapse experience: patient-reported outcomes from the North American Research Committee on Multiple Sclerosis (NARCOMS) Registry. BMC Neurol. 2013 Sep 10;13:119. doi: 10.1186/1471-2377-13-119. PMID 24016260
- [Background] Hirst C, Ingram G, Pearson O, Pickersgill T, Scolding N, Robertson N. Contribution of relapses to disability in multiple sclerosis. J Neurol. 2008 Feb;255(2):280-7. doi: 10.1007/s00415-008-0743-8. Epub 2008 Jan 23. PMID 18204919
- [Background] Lublin FD, Baier M, Cutter G. Effect of relapses on development of residual deficit in multiple sclerosis. Neurology. 2003 Dec 9;61(11):1528-32. doi: 10.1212/01.wnl.0000096175.39831.21. PMID 14663037
- [Background] Kwon S, Hermayer KL, Hermayer K. Glucocorticoid-induced hyperglycemia. Am J Med Sci. 2013 Apr;345(4):274-277. doi: 10.1097/MAJ.0b013e31828a6a01. PMID 23531958
- [Background] Johnston KC, Hall CE, Kissela BM, Bleck TP, Conaway MR; GRASP Investigators. Glucose Regulation in Acute Stroke Patients (GRASP) trial: a randomized pilot trial. Stroke. 2009 Dec;40(12):3804-9. doi: 10.1161/STROKEAHA.109.561498. Epub 2009 Oct 15. PMID 19834016
- [Background] Baker L, Juneja R, Bruno A. Management of hyperglycemia in acute ischemic stroke. Curr Treat Options Neurol. 2011 Dec;13(6):616-28. doi: 10.1007/s11940-011-0143-8. PMID 21861124
- [Background] Southerland AM, Johnston KC. Considering hyperglycemia and thrombolysis in the Stroke Hyperglycemia Insulin Network Effort (SHINE) trial. Ann N Y Acad Sci. 2012 Sep;1268(1):72-8. doi: 10.1111/j.1749-6632.2012.06731.x. PMID 22994224
- [Background] Bruno A, Biller J, Adams HP Jr, Clarke WR, Woolson RF, Williams LS, Hansen MD. Acute blood glucose level and outcome from ischemic stroke. Trial of ORG 10172 in Acute Stroke Treatment (TOAST) Investigators. Neurology. 1999 Jan 15;52(2):280-4. doi: 10.1212/wnl.52.2.280. PMID 9932944
- [Background] Fang Y, Zhang S, Wu B, Liu M. Hyperglycaemia in acute lacunar stroke: a Chinese hospital-based study. Diab Vasc Dis Res. 2013 May;10(3):216-21. doi: 10.1177/1479164112459663. Epub 2012 Oct 18. PMID 23079541
- [Background] Matute C, Domercq M, Perez-Samartin A, Ransom BR. Protecting white matter from stroke injury. Stroke. 2013 Apr;44(4):1204-11. doi: 10.1161/STROKEAHA.112.658328. Epub 2012 Dec 4. No abstract available. PMID 23212168
- [Background] Wens I, Dalgas U, Deckx N, Cools N, Eijnde BO. Does multiple sclerosis affect glucose tolerance? Mult Scler. 2014 Aug;20(9):1273-6. doi: 10.1177/1352458513515957. Epub 2013 Dec 17. PMID 24347183
- [Background] Sternberg Z, Leung C, Sternberg D, Li F, Karmon Y, Chadha K, Levy E. The prevalence of the classical and non-classical cardiovascular risk factors in multiple sclerosis patients. CNS Neurol Disord Drug Targets. 2013 Feb 1;12(1):104-11. doi: 10.2174/1871527311312010016. PMID 23244431
- [Background] Marrie RA, Rudick R, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. Vascular comorbidity is associated with more rapid disability progression in multiple sclerosis. Neurology. 2010 Mar 30;74(13):1041-7. doi: 10.1212/WNL.0b013e3181d6b125. PMID 20350978
- [Background] Marrie RA, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. Comorbidity delays diagnosis and increases disability at diagnosis in MS. Neurology. 2009 Jan 13;72(2):117-24. doi: 10.1212/01.wnl.0000333252.78173.5f. Epub 2008 Oct 29. PMID 18971448
- [Background] Sellebjerg F, Frederiksen JL, Nielsen PM, Olesen J. Double-blind, randomized, placebo-controlled study of oral, high-dose methylprednisolone in attacks of MS. Neurology. 1998 Aug;51(2):529-34. doi: 10.1212/wnl.51.2.529. PMID 9710030
- [Background] Eriksson M, Andersen O, Runmarker B. Long-term follow up of patients with clinically isolated syndromes, relapsing-remitting and secondary progressive multiple sclerosis. Mult Scler. 2003 Jun;9(3):260-74. doi: 10.1191/1352458503ms914oa. PMID 12814173
- [Background] Langer-Gould A, Popat RA, Huang SM, Cobb K, Fontoura P, Gould MK, Nelson LM. Clinical and demographic predictors of long-term disability in patients with relapsing-remitting multiple sclerosis: a systematic review. Arch Neurol. 2006 Dec;63(12):1686-91. doi: 10.1001/archneur.63.12.1686. PMID 17172607
- [Background] Marrie RA, Horwitz R, Cutter G, Tyry T. Cumulative impact of comorbidity on quality of life in MS. Acta Neurol Scand. 2012 Mar;125(3):180-6. doi: 10.1111/j.1600-0404.2011.01526.x. Epub 2011 May 26. PMID 21615355
- [Background] Godoy DA, Di Napoli M, Rabinstein AA. Treating hyperglycemia in neurocritical patients: benefits and perils. Neurocrit Care. 2010 Dec;13(3):425-38. doi: 10.1007/s12028-010-9404-8. PMID 20652767
- [Background] Sala F, Menna G, Bricolo A, Young W. Role of glycemia in acute spinal cord injury. Data from a rat experimental model and clinical experience. Ann N Y Acad Sci. 1999;890:133-54. doi: 10.1111/j.1749-6632.1999.tb07989.x. PMID 10668421
- [Background] Zhao QJ, Zhang XG, Wang LX. Mild hypothermia therapy reduces blood glucose and lactate and improves neurologic outcomes in patients with severe traumatic brain injury. J Crit Care. 2011 Jun;26(3):311-5. doi: 10.1016/j.jcrc.2010.08.014. Epub 2010 Oct 2. PMID 20889287
- [Background] Selwyn R, Hockenbury N, Jaiswal S, Mathur S, Armstrong RC, Byrnes KR. Mild traumatic brain injury results in depressed cerebral glucose uptake: An (18)FDG PET study. J Neurotrauma. 2013 Dec 1;30(23):1943-53. doi: 10.1089/neu.2013.2928. Epub 2013 Oct 2. PMID 23829400
- [Background] Johnston KC, Connors AF Jr, Wagner DP, Knaus WA, Wang X, Haley EC Jr. A predictive risk model for outcomes of ischemic stroke. Stroke. 2000 Feb;31(2):448-55. doi: 10.1161/01.str.31.2.448. PMID 10657421
- [Background] Hacke W, Donnan G, Fieschi C, Kaste M, von Kummer R, Broderick JP, Brott T, Frankel M, Grotta JC, Haley EC Jr, Kwiatkowski T, Levine SR, Lewandowski C, Lu M, Lyden P, Marler JR, Patel S, Tilley BC, Albers G, Bluhmki E, Wilhelm M, Hamilton S; ATLANTIS Trials Investigators; ECASS Trials Investigators; NINDS rt-PA Study Group Investigators. Association of outcome with early stroke treatment: pooled analysis of ATLANTIS, ECASS, and NINDS rt-PA stroke trials. Lancet. 2004 Mar 6;363(9411):768-74. doi: 10.1016/S0140-6736(04)15692-4. PMID 15016487
- [Background] Vespa P, McArthur DL, Stein N, Huang SC, Shao W, Filippou M, Etchepare M, Glenn T, Hovda DA. Tight glycemic control increases metabolic distress in traumatic brain injury: a randomized controlled within-subjects trial. Crit Care Med. 2012 Jun;40(6):1923-9. doi: 10.1097/CCM.0b013e31824e0fcc. PMID 22610193
- [Background] Moro N, Ghavim S, Harris NG, Hovda DA, Sutton RL. Glucose administration after traumatic brain injury improves cerebral metabolism and reduces secondary neuronal injury. Brain Res. 2013 Oct 16;1535:124-36. doi: 10.1016/j.brainres.2013.08.044. Epub 2013 Aug 29. PMID 23994447
- [Background] Nijland PG, Michailidou I, Witte ME, Mizee MR, van der Pol SM, van Het Hof B, Reijerkerk A, Pellerin L, van der Valk P, de Vries HE, van Horssen J. Cellular distribution of glucose and monocarboxylate transporters in human brain white matter and multiple sclerosis lesions. Glia. 2014 Jul;62(7):1125-41. doi: 10.1002/glia.22667. Epub 2014 Apr 1. PMID 24692237
- [Background] Bruno A, Kent TA, Coull BM, Shankar RR, Saha C, Becker KJ, Kissela BM, Williams LS. Treatment of hyperglycemia in ischemic stroke (THIS): a randomized pilot trial. Stroke. 2008 Feb;39(2):384-9. doi: 10.1161/STROKEAHA.107.493544. Epub 2007 Dec 20. PMID 18096840
- [Background] Pulsinelli WA, Levy DE, Sigsbee B, Scherer P, Plum F. Increased damage after ischemic stroke in patients with hyperglycemia with or without established diabetes mellitus. Am J Med. 1983 Apr;74(4):540-4. doi: 10.1016/0002-9343(83)91007-0. PMID 6837584
- [Background] Lassmann H. Hypoxia-like tissue injury as a component of multiple sclerosis lesions. J Neurol Sci. 2003 Feb 15;206(2):187-91. doi: 10.1016/s0022-510x(02)00421-5. PMID 12559509
- [Background] Zivadinov R, Rudick RA, De Masi R, Nasuelli D, Ukmar M, Pozzi-Mucelli RS, Grop A, Cazzato G, Zorzon M. Effects of IV methylprednisolone on brain atrophy in relapsing-remitting MS. Neurology. 2001 Oct 9;57(7):1239-47. doi: 10.1212/wnl.57.7.1239. PMID 11591843
- [Background] Viardot A, Grey ST, Mackay F, Chisholm D. Potential antiinflammatory role of insulin via the preferential polarization of effector T cells toward a T helper 2 phenotype. Endocrinology. 2007 Jan;148(1):346-53. doi: 10.1210/en.2006-0686. Epub 2006 Sep 28. PMID 17008395
- [Background] Wieser V, Moschen AR, Tilg H. Inflammation, cytokines and insulin resistance: a clinical perspective. Arch Immunol Ther Exp (Warsz). 2013 Apr;61(2):119-25. doi: 10.1007/s00005-012-0210-1. Epub 2013 Jan 10. PMID 23307037
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Kallaur AP, Oliveira SR, Colado Simao AN, Delicato de Almeida ER, Kaminami Morimoto H, Lopes J, de Carvalho Jennings Pereira WL, Marques Andrade R, Muliterno Pelegrino L, Donizete Borelli S, Kaimen-Maciel DR, Reiche EM. Cytokine profile in relapsing-remitting multiple sclerosis patients and the association between progression and activity of the disease. Mol Med Rep. 2013 Mar;7(3):1010-20. doi: 10.3892/mmr.2013.1256. Epub 2013 Jan 2. PMID 23292766
- [Background] Rudick RA, Ransohoff RM. Cytokine secretion by multiple sclerosis monocytes. Relationship to disease activity. Arch Neurol. 1992 Mar;49(3):265-70. doi: 10.1001/archneur.1992.00530270079022. PMID 1536629
- [Background] Khalili M, Azimi A, Izadi V, Eghtesadi S, Mirshafiey A, Sahraian MA, Motevalian A, Norouzi A, Sanoobar M, Eskandari G, Farhoudi M, Amani F. Does lipoic acid consumption affect the cytokine profile in multiple sclerosis patients: a double-blind, placebo-controlled, randomized clinical trial. Neuroimmunomodulation. 2014;21(6):291-6. doi: 10.1159/000356145. Epub 2014 May 6. PMID 24821457
- [Background] Imitola J, Chitnis T, Khoury SJ. Cytokines in multiple sclerosis: from bench to bedside. Pharmacol Ther. 2005 May;106(2):163-77. doi: 10.1016/j.pharmthera.2004.11.007. Epub 2005 Jan 11. PMID 15866318
- [Background] Schneider A, Long SA, Cerosaletti K, Ni CT, Samuels P, Kita M, Buckner JH. In active relapsing-remitting multiple sclerosis, effector T cell resistance to adaptive T(regs) involves IL-6-mediated signaling. Sci Transl Med. 2013 Jan 30;5(170):170ra15. doi: 10.1126/scitranslmed.3004970. PMID 23363979
- [Background] Warabi Y. Role of IL-1 and potential therapies in multiple sclerosis. Drug Discovery Today: Therapeutic Strategies 2007;4:19-24.
- [Background] Juhler M. Simultaneous determination of regional cerebral blood flow, glucose metabolism, and pH in acute experimental allergic encephalomyelitis. J Cereb Blood Flow Metab. 1987 Oct;7(5):578-84. doi: 10.1038/jcbfm.1987.108. PMID 3654798
- [Background] Juhler M. Pathophysiological aspects of acute experimental allergic encephalomyelitis. Acta Neurol Scand Suppl. 1988;119:1-21. doi: 10.1111/j.1600-0404.1988.tb08016.x. PMID 3064529
- [Background] JONES HH, JONES HH Jr, BUNCH LD. Biochemical studies in multiple sclerosis. Ann Intern Med. 1950 Oct;33(4):831-40. doi: 10.7326/0003-4819-33-4-831. No abstract available. PMID 14771754
- [Background] Sternberg Z, Leung C, Sternberg D, Yu J, Hojnacki D. Disease modifying therapies modulate cardiovascular risk factors in patients with multiple sclerosis. Cardiovasc Ther. 2014 Apr;32(2):33-9. doi: 10.1111/1755-5922.12049. PMID 24119301
- [Background] Mowry EM, Pesic M, Grimes B, Deen S, Bacchetti P, Waubant E. Demyelinating events in early multiple sclerosis have inherent severity and recovery. Neurology. 2009 Feb 17;72(7):602-8. doi: 10.1212/01.wnl.0000342458.39625.91. PMID 19221292
- [Background] Penesova A, Vlcek M, Imrich R, Vernerova L, Marko A, Meskova M, Grunnerova L, Turcani P, Jezova D, Kollar B. Hyperinsulinemia in newly diagnosed patients with multiple sclerosis. Metab Brain Dis. 2015 Aug;30(4):895-901. doi: 10.1007/s11011-015-9665-1. Epub 2015 Mar 27. PMID 25809135
- [Background] SCHUMACHER GA, BEEBE G, KIBLER RF, KURLAND LT, KURTZKE JF, MCDOWELL F, NAGLER B, SIBLEY WA, TOURTELLOTTE WW, WILLMON TL. PROBLEMS OF EXPERIMENTAL TRIALS OF THERAPY IN MULTIPLE SCLEROSIS: REPORT BY THE PANEL ON THE EVALUATION OF EXPERIMENTAL TRIALS OF THERAPY IN MULTIPLE SCLEROSIS. Ann N Y Acad Sci. 1965 Mar 31;122:552-68. doi: 10.1111/j.1749-6632.1965.tb20235.x. No abstract available. PMID 14313512